CLINICAL TRIAL: NCT05887388
Title: Adapting Connect-Home Transitional Care to Fit the Unique Needs of Persons With Alzheimer's Disease and Other Dementias and Their Caregivers: A Pilot Study
Brief Title: Adapting Connect-Home Transitional Care for the Unique Needs of Persons With Alzheimer's Disease and Other Dementias and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-2406; R01NR017636-03 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Pathologic Processes
Keywords: Transitional Care; Skilled Nursing Facilities
MeSH Terms: conditions — Pathologic Processes

STUDY DESIGN:
Intervention Model Description: This feasibility and acceptability study will use a single-arm, post-test-only trial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Connect-Home Plus will be delivered in the skilled nursing facility and via telephone after discharge.
  Interventions: Behavioral: Connect-Home Plus

INTERVENTIONS:
Behavioral: Connect-Home Plus — Connect-Home Plus will introduce organizational structure to support delivery of transitional care processes. New elements of structure include:electronic health record (EHR) template, Connect-Home Plus Toolkit, and Staff Training. After structural elements are added, SNF staff will use Connect-Home Plus care processes to deliver the 2-step transitional care intervention.In Step 1, SNF nurses,therapists, and social workers will develop a Transition Plan of Care and prepare the patient and caregiver to manage the illness and functional needs. In Step 2, a dementia caregiving specialist will call the patient's home three times within 30 days of discharge. Both intervention steps will focus on key care needs, such as 1) home safety; 2) care of symptoms of ADRD; 3) symptom management; 4) medication reconciliation; 5) function and activity; and 6) coordination of follow-up medical care.

SUMMARY:
This primary purpose of this study will be to (1) examine the feasibility and acceptability of transitional care focusing on care needs of skilled nursing facility (SNF) patients with dementia and their caregivers (primary aim). The secondary purpose will be to describe the effect of the intervention on SNF patient outcomes (preparedness for discharge, quality of life, function and acute care use) and caregiver outcomes (preparedness for the caregiving role, caregiver burden and caregiver distress).

DETAILED DESCRIPTION:
Persons with Alzheimer's disease and related dementia (ADRD) and their caregivers confront complex health challenges during transfers from skilled nursing facilities (SNF) to home, such as recent acute illness and functional losses, incurable medical conditions, patient dependence on family caregivers, and sequelae of declining cognitive ability, such as agitated or aggressive behavior and depression. Other research indicates that usual discharge planning does not address the unique care needs of SNF patients with ADRD and caregiver dyads as they prepare for SNF discharge and begin home-based care. Building on our previous studies and observational studies of unmet care needs of SNF patients with ADRD and their caregivers, the investigators developed Connect-Home Plus, a transitional care intervention to prepare dyads for SNF discharge and caregiver support at home after SNF discharge.

Connect-Home Plus will provide new versions of the Connect-Home transitional plan of care EHR template, toolkit, and staff training protocol. The adapted version will support staff in tailoring the transitional care processes to fit the needs of persons with ADRD and their caregivers. It will include (1) new tools to move staff stepwise through a process to prepare persons with AD/ADRD for discharge, and (2) staff training to increase the ability of staff to tailor transitional care plans for the unique needs of persons with ADRD and their caregivers.

The investigators will use a single-arm post-test-only trial design with a sample of 20 persons with ADRD and 20 caregivers in 2 SNFs over 6 months. The investigators will determine the feasibility and acceptability of Connect-Home Plus and estimated mean outcomes of persons with ADRD and their caregivers. Feasibility will be assessed with a chart review of SNF medical records. Acceptability will be assessed with questionnaire with patients and caregivers in 21 days after patient discharge from the SNF to home. Patient and caregiver outcomes will be assessed with questionnaires in 30 days after patient discharge from the SNF to home. Data will be analyzed using descriptive statistics.

ELIGIBILITY:
Patient Inclusion Criteria:

* be able to speak English
* have a goal of discharge to home
* have a diagnosis of ADRD, or a Brief Inventory of Mental Status (BIMS) score <13, or (for persons unable to complete the BIMS assessment), have a Cognitive performance score of ≥3 (calculated using data in the Minimum Data Set 3.0 and an algorithm for estimating cognitive impairment using Minimum Data Set 3.0 data other than BIMS)
* have a caregiver willing to participate.
* for patients with documentation in the medical record of a caregiver who is the patient's legally authorized representative, consent of the caregiver to participate in the study as the patient's representative.

Patient Exclusion Criteria:

* unable to speak English

Caregiver Inclusion Criteria

* self-reports assisting the patient at home
* the ability to speak English.

Caregiver Exclusion Criteria

* unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Toles, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigators who propose to use the data must have approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Connect-Home Plus will be delivered in the skilled nursing facility (SNF) and via telephone after discharge.
  Connect-Home Plus: Connect-Home Plus will introduce organizational structure to support delivery of transitional care processes. New elements of structure include:electronic health record (EHR) template, Connect-Home Plus Toolkit, and Staff Training. After structural elements are added, SNF staff will use Connect-Home Plus care processes to deliver the 2-step transitional care intervention.In Step 1, SNF nurses,therapists, and social workers will develop a Transition Plan of Care and prepare the patient and caregiver to manage the illness and functional needs. In Step 2, a home health care nurse will visit (one time) and a dementia caregiving specialist will call the patient's home three times within 30 days of discharge. Both intervention steps will focus on key care needs, such as 1) home safety; 2) care of symptoms of Alzheimer's disease and related dementia (ADRD); 3) symptom management; 4) medication reconciliation; 5) function and activity; and 6) coordination of follow-up medical care.
Period: Overall Study
Arm/Group | Intervention
Started | 38
Patients Started | 19
Caregivers Started | 19
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for Patients and Caregivers.
  years
    Patients: number analyzed (Participants) | 19
    Patients | 85.4 (6.8)
    Caregivers: number analyzed (Participants) | 19
    Caregivers | 61.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 19
    Patients: Female | 15
    Patients: Male | 4
    Caregivers: number analyzed (Participants) | 19
    Caregivers: Female | 13
    Caregivers: Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 19
    Patients: Hispanic or Latino | 0
    Patients: Not Hispanic or Latino | 19
    Patients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 19
    Caregivers: Hispanic or Latino | 0
    Caregivers: Not Hispanic or Latino | 19
    Caregivers: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 19
    Patients: American Indian or Alaska Native | 0
    Patients: Asian | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0
    Patients: Black or African American | 1
    Patients: White | 18
    Patients: More than one race | 0
    Patients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 19
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 1
    Caregivers: White | 18
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Patients | 19
  United States: Caregivers | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients for Whom the Intervention Components Were Feasible
Description: Feasibility will measured using an instrument to audit skilled nursing facility medical records of the patient and the intervention log of services for the Patient and Caregiver dyad. It includes eight dichotomous (yes-no) items that indicate feasibility of the Connect-Home Plus intervention. The feasibility items include: (1) completing the Transition Plan of Care; (2) convening the care plan meeting with caregiver attending; (3) reviewing advance directives in the SNF; (4) scheduling follow-up medical appointments; (5) transmitting records to follow-up clinicians; (6) home care nurse completion of the first home visit within 24 hours after discharge; (7) completion of first caregiver support call within 72 hours of discharge; (8) completion of the second and third caregiver support call within one month of discharge. A "Yes" answer indicates that the intervention component was feasible to provide for the patient and caregiver dyad.
Time Frame: 30 days after SNF discharge
Population: Data are reported only for Patients as this measure does not apply to Caregivers.
Measure: Count of Participants; unit: Participants
Groups:
- Connect-Home Plus Patients: Connect-Home Plus will be delivered in the skilled nursing facility and via telephone after discharge.
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 19
Participants
  Transition Plan of Care | 16
  Care plan meeting | 19
  Advance directives | 15
  Follow-up medical appointments | 16
  Record transmission | 19
  Home visit within 24 hours | 17
  Call back #1 within 72 hours | 17
  Call back #2 and #3 within 30 days | 16

2. Primary Outcome: Mean Patient Intervention Satisfaction Scores
Description: This interview guide will be used to assess the acceptability of Connect-Home Plus with persons with ADRD. The interview will include questions about (1) factors that made the Connect-Home Plus transitional care services easy or difficult to use, (2) specific supports that were and were not helpful, (3) the effect of Connect-Home Plus on how to manage issues related to ADRD at home, and (4) unmet needs for care of issues related to ADRD at home. Responses to the interview guide questions will be used to generate 3 4-point Likert scale acceptability scores, including (1) how helpful was Connect-Home Plus, (2) how difficult were these services to use, and (3) how well did these services prepare you for care at home. The scores will include 0 meaning not applicable, and scores 1-3 indicating acceptability, with lower scores indicating higher acceptability.
Time Frame: 21 days after SNF discharge
Population: Data are reported only for Patients as this measure does not apply to Caregivers. Fifteen Patients were unable or unavailable to participate in data collection for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 4
score on a scale
  Helpfulness | 1.0 (0)
  Usefulness | 1.0 (0)
  Appropriateness | 1.0 (0)

3. Primary Outcome: Mean Caregiver Intervention Satisfaction Scores
Description: This interview guide will be used to assess the acceptability of Connect-Home Plus with caregivers of persons with ADRD. This interview guide will include questions about (1) factors that made the Connect-Home Plus transitional care services easy or difficult to use, (2) specific supports that were and were not helpful, (3) the effect of Connect-Home Plus on how to manage issues related to ADRD at home, and (4) unmet needs for care of issues related to ADRD at home. Responses to the interview guide questions will be used to generate 3 4-point Likert scale acceptability scores, including (1) how helpful was Connect-Home Plus, (2) how difficult were these services to use, and (3) how well did these services prepare you for care at home. The scores will include 0 meaning not applicable, and scores 1-3 indicating acceptability, with lower scores indicating higher acceptability
Time Frame: 21 days after SNF discharge
Population: Data are reported only for Caregivers as this measure does not apply to Patients. Seven Caregivers were unavailable to participate in data collection for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Connect-Home Plus Caregivers: Connect-Home Plus will be delivered in the skilled nursing facility and via telephone after discharge.
Arm/Group | Connect-Home Plus Caregivers
Number analyzed (Participants) | 12
score on a scale
  Helpfulness | 1.3 (0.5)
  Usefulness | 1.0 (0)
  Appropriateness | 1.3 (0.5)

4. Secondary Outcome: Care Transitions Measure-15 (Patient)
Description: The patient's preparedness for discharge will be measured by the Care Transitions Measure-15 (CTM-15), which includes 15 items on a 4-point scale. The CTM-15 measures self-reported knowledge and skills for continuing care at home. Summary scores range 0-100, with higher scores indicating greater preparedness. Data collected from either the Patient or the Caregiver serving as proxy.
Time Frame: 7 Days After SNF Discharge
Population: Data are reported only for Patients as this measure does not apply to Caregivers and data are reported by the Patient (or the Caregiver serving as a proxy). Participants were unavailable for data collection for 3 Patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 16
score on a scale | 70.3 (12.0)

5. Secondary Outcome: Preparedness for Caregiving Scale (Caregiver)
Description: The caregiver's preparedness for caregiving will be measured by the Preparedness for Caregiving Scale (PCS), which includes 8 items on a five-point Likert scale (0-4). The PCS measures self-reported readiness for caregiving. Range = 0-32, with higher scores associated with greater preparedness.
Time Frame: 7 Days After SNF Discharge
Population: Data are reported only for Caregivers as this measure does not apply to Patients. Three Caregivers were unavailable for data collection for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Caregivers
Number analyzed (Participants) | 16
score on a scale | 24.8 (12.4)

6. Secondary Outcome: Life Space Assessment
Description: Patient's function will be measured using the Life Space Assessment, which includes 5 Likert scales corresponding to a hierarchy of levels of mobility (each scored from 0-4) where weights are the product of the "Life-space level" (range 1-5) and the"independence" score (range 1-2). The range is 1-120. Lower scores are associated with less life-space.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for Patients as this measure does not apply to Caregivers and data are reported by the Patient (or the Caregiver serving as a proxy). Participants were unavailable for data collection for 5 Patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 14
score on a scale | 20.1 (9.6)

7. Secondary Outcome: Dementia Quality of Life Measure (Patient)
Description: The quality of life of the person with ADRD will be assessed with the Dementia Quality of Life Measure. It has 28 items that cover four quality of life dimensions: daily activities, memory, negative emotion and positive emotion. The score range is 28-112 with higher scores indicating better quality of life.
Time Frame: 30 Days After SNF Discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 4
score on a scale | 90.8 (9.9)

8. Secondary Outcome: Dementia Quality of Life-Proxy Measure (Caregiver)
Description: When the Patient was unable to answer the DEMQOL, the Caregiver was surveyed with the DEMQOL-Proxy. With this measure, the score range is 31-124 with higher scores indicating better quality of life.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for Caregivers as this measure does not apply to Patients. Four Patients reported DEMQOL themselves (and thus did not need proxy report) and 5 Caregivers were unavailable for data collection with this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Caregivers
Number analyzed (Participants) | 10
score on a scale | 91.1 (10.3)

9. Secondary Outcome: Mean Self-Reported Days of ED or Hospital Use 30 Days After Skilled Nursing Facility Discharge (Patient)
Description: Patient's days of acute care use will be measured using the self-reported number of combined number of days the patients pends in the Emergency Department (ED) or hospital in 30 days after SNF discharge.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for Patients as this measure does not apply to Caregivers and data are reported by the Patient (or the Caregiver serving as a proxy).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Connect-Home Plus Patients
Number analyzed (Participants) | 19
days | 0.58 (1.7)

10. Secondary Outcome: Zarit Caregiver Burden Scale (Caregiver)
Description: Caregiver burden will be measured using the Zarit Caregiver Burden Scale, which includes 12 items on a five-point scale,measuring caregiver perceptions that "caregiving has an adverse effect on their emotional, social, financial, physical and spiritual functioning." Scores range 0-48; higher scores are associated with greater burden.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for Caregivers as this measure does not apply to Patients. Five Caregivers were unavailable for data collection for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Caregivers
Number analyzed (Participants) | 14
score on a scale | 16.6 (6.6)

11. Secondary Outcome: Distress Thermometer (Caregiver)
Description: Caregiver distress will be measured using the Distress Thermometer, which includes 1 item on an 11-point scale, measuring negative affect (e.g., sadness and fear) related to caregiving for a severely ill person. Score ranges 0-10, with scores >4 associated with distress.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for Caregivers as this measure does not apply to Patients. Five Caregivers were unavailable to participate in data collection for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home Plus Caregivers
Number analyzed (Participants) | 14
score on a scale | 4.1 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from when participants entered the study to when they completed study procedures, an approximate total of up to 60 days.
Description: Due to the severity of illness present in the study population, unrelated adverse events were expected during this study.
Groups:
- Patients; Caregivers: Connect-Home Plus will be delivered in the skilled nursing facility and via telephone after discharge.
  Connect-Home Plus: Connect-Home Plus will introduce organizational structure to support delivery of transitional care processes. New elements of structure include:electronic health record (EHR) template, Connect-Home Plus Toolkit, and Staff Training. After structural elements are added, SNF staff will use Connect-Home Plus care processes to deliver the 2-step transitional care intervention.In Step 1, SNF nurses,therapists, and social workers will develop a Transition Plan of Care and prepare the patient and caregiver to manage the illness and functional needs. In Step 2, a home health care nurse will visit (one time) and a dementia caregiving specialist will call the patient's home three times within 30 days of discharge. Both intervention steps will focus on key care needs, such as 1) home safety; 2) care of symptoms of ADRD; 3) symptom management; 4) medication reconciliation; 5) function and activity; and 6) coordination of follow-up medical care.
Arm/Group | Patients | Caregivers
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=19) | Caregivers (N=19)
Acute UTI (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT05887388/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05887388/ICF_001.pdf